# Document Cover Page

# **Consent Form**

# **Study Title:**

Promoting Protection of Others to Increase Future COVID-19 Booster Shot Vaccination Intentions in Younger Adult Canadians: Evaluating the Efficacy of Short Video-based Interventions

NCT number: Not assigned

**Date of Document:** February 27th 2023


Centre intégré
universitaire de santé
et de services sociaux
du Centre-Ouestde-l'Île-de-Montréal

Québec

Hôpital général juif
Jewish General Hospital

INSTITUTE OF COMMUNITY AND FAMILY PSYCHIATRY 4333, CÔTE SAINTE-CATHERINE ROAD, MONTREAL, QC, H3T 1E4

UTILISATION ADMINISTRATIVE UNIQUEMENT PAR LE CER

**SITE:** Lady Davis Institute for Medical Research, Jewish General Hospital

**Department:** Psychosocial Research **Lead Investigator:** Zeev Rosberger

Co-Investigators : Gregory Zimet (Indiana University), Matthew Tunis (Public Health Agency of

Canada), Ève Dubé (Quebec National Institute of Public Health), Ovidiu Tatar, Samara Perez

Funding source: Canadian Institutes of Health Research (CIHR)

#### INFORMATION AND CONSENT FORM

**Research project title:** Exploring the effect of a video intervention on COVID-19 vaccination intentions

## INTRODUCTION

You are invited to participate in a research project. This research is being conducted to study the effect of different health messages related to COVID-19 vaccination. You are being asked to participate in this research because you are a young adult (aged 18-39) who may be eligible for COVID-19 vaccination. To make an informed decision, you have the right to know the purpose and procedures used in this research as well as the potential benefits, risks, disadvantages, and compensation associated with it.

Before agreeing to participate in this research project, please read the information contained in this consent form. We encourage you to ask the researcher responsible for this research project or a member of the research team as many questions as you feel are necessary to understand the implications of your participation (see contact information below). You do not have to participate in this research project if you do not wish to.

If you decide to participate in the project, you will be asked to select "Continue" below.

#### NATURE AND OBJECTIVES OF THE RESEARCH PROJECT

This study aims to evaluate different messages related to the COVID-19 vaccine for young adults. Your answers will be helpful in deciding how to communicate with the Canadian public about


COVID-19 vaccination in the future. The project is led by Dr. Zeev Rosberger's lab at the Lady Davis Institute for Medical Research.

## CONDUCT OF THE RESEARCH PROJECT

This survey should take about 15 minutes. As part of this survey, you will be randomly assigned to watch one of three videos related to COVID-19 vaccination. You will also be asked questions about yourself, your health behaviours, and your attitudes towards COVID-19 and vaccination.

### RISKS AND DISADVANTAGES OF PARTICIPATING IN RESEARCH

Participating in this research study carries no known or serious risks. Some questions asked during the research process may cause you distress or other negative emotions. If you feel discomfort, you are free to stop at any time.

If you feel discomfort as result of the survey, you can access mental health support in your area through the resources available on the government's webpage:

https://www.canada.ca/en/public-health/topics/mental-health-wellness.html

Information about you will be collected electronically, using devices, applications, and tools for transferring and storing data over the internet. The researcher responsible for this research is committed to protecting your personal data (see "confidentiality" section below) and the collection of data is completely confidential.

## POTENTIAL BENEFITS OF PARTICIPATING IN RESEARCH

You will not receive any direct personal benefit from your participation in this study, but we hope that the research findings will contribute to the development of policies and messages to reduce transmission, hospitalizations and deaths related to the COVID-19 virus.

For more information on COVID-19 vaccines, you can visit the websites listed at the end of the survey.

#### **DECLARATION OF CONFLICT OF INTEREST**

The researcher responsible for this research has no conflicts of interest to declare.

## PLANNED COMPENSATION

[IF DYNATA PANELIST SHOW:] You will be compensated for completing this survey according to the terms of Dynata's rewards program (see section 8 of the Dynata terms and conditions). You may have the opportunity to accumulate rewards, incentives and entries into prize draws or sweepstakes. Incentives may be in the form of points or dollars. Information, official rules and terms and conditions for rewards, incentives and prize draws or sweepstakes may be available in Dynata's terms and conditions, on the website for a panel, at the beginning or end of a survey, in survey invitations, on the website(s) or webpage(s) for redeeming rewards, incentives, and prizes,


and/or may be described in any newsletter or other communication distributed or published by Dynata.

[IF OTHER CANADIAN PARTICIPANT SHOW:] You will be compensated for completing this survey according to the terms of your panel's rewards program.

#### CONFIDENTIALITY

The Principal Investigator is responsible for the confidentiality and security of research data.

During your participation in this research project, the researcher responsible for the project and the research team will collect, in a research file, the information about you that is necessary to meet the scientific objectives of the research project. This information includes personally identifiable information (biological sex, gender, age, ethnicity, education, occupation) and the information provided in this questionnaire.

All information collected as part of this research project will be collected anonymously and will remain confidential. This data will be stored on a secure password-protected file share on the server of the Lady Davis Institute for Medical Research, CIUSSS West-Central Montreal for 10 years. The principal investigator, Dr. Zeev Rosberger, is responsible for the data. By completing this online survey, your identity will not be known to the research team. Dynata only uses sociodemographic identifying information to recruit eligible participants based on our research criteria and collects your Participant ID and IP address to prevent you repeating the survey. IP addresses are not retained after the completion of the project. None of this information is shared with the research team. Dynata will send anonymous survey data to the research team.

# **VOLUNTARY PARTICIPATION AND RIGHT OF WITHDRAWAL**

Your participation in this research project is voluntary and ongoing. You are free to refuse to participate. You can withdraw from this search at any time, without having to give reasons. If you withdraw from the research project, no further data will be collected. Data already collected as part of this research will nevertheless be retained, analyzed, or used to ensure the integrity of the research project, as specified in this document.

# FUTURE USE OF DATA, COMMUNICATION AND PUBLICATION OF RESEARCH RESULTS

Results may be published in academic journals, presented at conferences, or discussed at knowledge exchange activities, but it will be impossible to identify you.

## **CONTACTS**

If you have any questions or problems related to the research project, or if you wish to withdraw from it, you may contact the lead investigator or a member of the research team: the lead investigator, Dr. Zeev Rosberger at (514) 340-8222 ext. 24215 or at zeev.rosberger@mcgill.ca or the study coordinator, Ben Haward to benjamin.haward@mail.mcgill.ca.

If you have any questions about your rights as a participant in this research project, or if you have any complaints or comments, please contact:


The Local Commissioner of Complaints and Quality of Services of the CIUSSS West-Central Montreal at (514) 340-8222 ext. 24222.

# STATEMENT OF ETHICAL APPROVAL

The CIUSSS West-Central Montreal REB Psychosocial Research Ethics Board (PSY) has given ethics approval to the research project and will monitor it.


# **SIGNATURE**

**Title:** Exploring the effect of a video intervention on COVID-19 vaccination intentions

I have read the information and consent form. By completing this questionnaire, it is understood that I do not waive my legal rights. My participation in this research is voluntary and I can withdraw from it at any time without consequence and without having to give reasons.

After reflection, I agree to participate in this research project under the conditions set out in this consent form.

If you agree to participate in this research, please select "continue"
